CLINICAL TRIAL: NCT01300026
Title: A Phase 1, First-in-Human Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 319 in Adult Subjects With Relapsed or Refractory Lymphoid Malignancies
Brief Title: AMG 319 Lymphoid Malignancy FIH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20101262; AMG 319 FIH Lymphoid
Record Dates: First submitted 2011-01-06; First posted 2011-02-21 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Cancer; Chronic Lymphocytic Leukemia; Diffuse Large Cell Lymphoma; Hematologic Malignancies; Hematology; Leukemia; Low Grade Lymphoma; Lymphoma; Mantle Cell Lymphoma; Non-Hodgkin's Lymphoma; Oncology; Oncology Patients; T Cell Lymphoma; Tumors
Keywords: Low intermediate grade B cell Lymphoma; Non-cutaneous T-cell NHL; Mantle Cell Lymphoma; PI3K delta; Lymphoid; NHL; MCL; Hematologic; CLL; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Hematologic Neoplasms; Leukemia; Lymphoma, Non-Hodgkin; Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, T-Cell | interventions — N-(1-(7-fluoro-2-(pyridin-2-yl)quinolin-3-yl)ethyl)-9H-purin-6-amine

ARMS (2):
- Part II Dose Expansion (Experimental): Dose selected from Part I dose exploration
  Interventions: Drug: AMG 319
- Part I Dose Exploration (Experimental): The AMG 319 doses proposed for this study are 25, 50, 100, 200, 300 and 400 mg administered by mouth once daily.
  Interventions: Drug: AMG 319

INTERVENTIONS:
Drug: AMG 319 — AMG 319 is a highly selective, orally bioavailable and potent small molecule inhibitor of PI3Kδ.

SUMMARY:
This is a multi-center, phase 1, open-label first-in-human study of AMG 319 in subjects with relapsed or refractory lymphoid malignancies. This study consists of two parts. The dose exploration in part 1, studies cohorts of 3 subjects with relapsed or refractory lymphoid malignancies and uses a practical continuous reassessment model [CRM] to guide dose escalation and to define the MTD. The dose expansion in part 2 will enroll 20 subjects with CLL at a dose no higher than the MTD and further explore the safety, PK, and clinical activity of AMG 319 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

- Part 1 (Dose Exploration): Relapsed or refractory lymphoid malignancy of the following type for which standard treatment does not exist or is no longer effective:

B-cell Chronic Lymphocytic Leukemia (CLL) confirmed by immunophenotype or Non-Hodgkin Lymphoma: Low or intermediate grade B-cell NHL, mantle cell lymphoma, non-cutaneous T-cell NHL confirmed by histology and/or immunophenotype

* Part 2 (Dose Expansion): Subjects must have relapsed or refractory B-cell Chronic Lymphocytic Leukemia confirmed by immunophenotype for which standard treatment does not exist or is no longer effective.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* Life expectancy of > 3 months, in the opinion of the investigator
* Men or women ≥ 18 years old
* Hematological function, as follows:

Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (unless due to disease-related bone marrow involvement as documented by bone marrow biopsy, ≥ 0.5 x 109/L) Platelet count ≥ 50 x 109/L (without a transfusion within 14 days before enrollment) Hemoglobin ≥ 9 g/dL

- Hepatic function, as follows: Aspartate aminotransferase (AST) < 3.0 x ULN Alanine aminotransferase (ALT) < 3.0 x ULN Alkaline phosphatase (ALP) < 2.0 x ULN (< 5 x ULN in subjects whom the PI and sponsor agree that clinical data suggest an extrahepatic source of elevation) Total bilirubin < 1.5 x ULN (< 3.0 x ULN for subjects with documented Gilbert's Disease or for whom the indirect bilirubin level suggests an extrahepatic source of elevation) Amylase ≤ 2.0 x IULN Lipase ≤ 2.0 x IULN

Exclusion Criteria:

* Primary or disseminated tumor involving the central nervous system (CNS)
* A history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer, or other solid tumors curatively treated with no evidence of disease for ≥ 2 years
* History of allogeneic stem-cell (or other organ) transplantation
* Clinically significant ECG changes which obscure the ability to assess the PR, QT, and QRS interval; congenital long QT syndrome
* QTcF interval > 470 msec
* Active or chronic hepatitis B or hepatitis C infection, determined by serologic tests
* Recent infection requiring intravenous anti-infective treatment that was completed ≤ 14 days before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-04; Primary Completion 2013-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Clinically significant or > or = to Grade 3 CTCAE changes in safety laboratory tests, physical exams, ECGs or vital signs | 28 Days after last subject enrolled per each cohort
PK parameters | 28 Days after last subject enrolled per each cohort
Clinical/radiological response rate for CLL subjects | With primary analysis
Treatment-emergent adverse events | 28 Days after last subject enrolled per each cohort

SECONDARY OUTCOMES:
Phospho-AKT level in circulating CLL cells | With primary analysis
Number of patients with clinical/radiological response | With primary analysis

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Research Site, Hackensack, New Jersey
  - Research Site, Durham, North Carolina
  - Research Site, Salt Lake City, Utah

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com